CLINICAL TRIAL: NCT05312931
Title: Retention of Knowledge and Skills of First Aid After Change in Concept of Teaching First Aid
Acronym: ReFA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Brno University Hospital (Other)
Responsible Party: Principal Investigator, Tereza Prokopova, MD, Principal investigator, Brno University Hospital
Other Study IDs: ReFA
Record Dates: First submitted 2022-02-17; First posted 2022-04-06 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: First Aid
Keywords: retention of knowledge; retention of skills; First Aid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: students who underwent original concept of First Aid
  Interventions: Other: OSCE
- Group B: student who underwent new concept of First Aid
  Interventions: Other: OSCE

INTERVENTIONS:
Other: OSCE — Students undergo OSCE (objective structured clinical exams). It means students will perform CPR for 2 min and their success rate will be monitored.

SUMMARY:
The investigators will evaluate the effect of simulation-based education in First Aid practice on knowledge and skills retention.

DETAILED DESCRIPTION:
In autumn semester 2020 a new concept of the subject First aid for the students of General medicine and Dentistry at Faculty of Medicine of Masaryk University was introduced. This concept based on evidence-based medical education puts different principles such as simulation-based education, learner-centred learning, peer learning and outcome-based education into practice.

First aid training (FAT) is indispensable part of the curriculum and knowledge of the first year medical students. The investigator´s aim is to evaluate if the new concept of the first aid training led to improvement in knowledge and mainly in skills of the students. Investigator´s null hypothesis is that the new concept does not lead to improvement in the long-term retention of the knowledge and the skills than the original concept. The investigators will compare tested knowledge and skills of the students who underwent FAT in autumn semester 2019 (original concept, group A) and the students who underwent FAT in autumn semester 2020 (new concept, group B).

The evaluation of the two groups will happen in the interval of 20-24 months after the completion of the FAT. Group A will be evaluated in autumn semester 2021, group B in autumn semester 2022. The evaluation method will be based on a knowledge test and a OSCE (objective structured clinical examination) stations.

Applying principles of evidence-based medical education into practice and designing FAT according to simulation-based education could lead better long-term retention of knowledge and skills of the students.

ELIGIBILITY:
Inclusion Criteria:

* Students of General medicine and Dentistry of the Faculty of Medicine of Masaryk University who underwent FAT in autumn semester 2020 and 2021 and have not been involved in Student as Teacher programme.

Exclusion Criteria:

* Students of General medicine and Dentistry of the Faculty of Medicine of Masaryk University who underwent FAT in different time intervals or who underwent FAT in autumn semester 2020 and 2021 and also have been involved in Student as Teacher programme.

Ages: 18 Years to 30 Years | Sex: All
Age Groups: Adult
Study Population: Students of General medicine and Dentistry of the Faculty of Medicine of Masaryk University who underwent FAT in autumn semester 2020 and 2021 and have not been involved in Student as Teacher programme.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Measurement of CPR quality - chest compression/ventilation ratio | Up to 36 months
  CPR quality will be measured with CPR monitoring (qCPR Anne - compression/ventilation feedback software). Attributes of CPR and a method of measurement:
  chest compression/ventilation ratio - investigator will count the number of chest compressions and a number of ventilation in each cycle in 2 min CPR. It will be statistically analyzed.
Measurement of CPR quality - percentage of adequate depth of chest compressions | Up to 36 months
  CPR quality will be measured with CPR monitoring (qCPR Anne - compression/ventilation feedback software). Attributes of CPR and a method of measurement:
  percentage of adequate depth of chest compressions (%) in 2 min CPR. Adequate depth of chest compression (5 - 6 cm).
  Method of mesurement: (qCPR Anne - compression/ventilation feedback software).
Measurement of CPR quality - the longest pause in chest compressions (s) | Up to 36 months
  CPR quality will be measured with CPR monitoring (qCPR Anne - compression/ventilation feedback software). Attributes of CPR and a method of measurement:
  the longest pause in chest compressions (s) in 2 min CPR. Method of mesurement: (qCPR Anne - compression/ventilation feedback software).
Measurement of CPR quality - percentage of chest compression when thorax was adequately released | Up to 36 months
  CPR quality will be measured with CPR monitoring (qCPR Anne - compression/ventilation feedback software). Attributes of CPR and a method of measurement:
  percentage of chest compression when thorax was adequately released (%) in 2 min CPR.
  Method of mesurement: (qCPR Anne - compression/ventilation feedback software).
Measurement of CPR quality - rescue breaths | Up to 36 months
  CPR quality will be measured with CPR monitoring (qCPR Anne - compression/ventilation feedback software). Attributes of CPR and a method of measurement:
  the number of detectable rescue breaths and number of unsuccessful rescue breaths during 2 min in CPR will be recorded. Detectable rescue breath means that the software was able to detect the rescue breath. Unsuccessful rescue breath means that the student tried to deliver rescue breath but the software was not able to detect it. Method of mesurement: (qCPR Anne - compression/ventilation feedback software).
Measurement of CPR quality - frequency of chest compressions | Up to 36 months
  CPR quality will be measured with CPR monitoring (qCPR Anne - compression/ventilation feedback software). Attributes of CPR and a method of measurement:
  frequency of chest compressions (compressions/min) in 2 min CPR will be measured with qCPR software. Method of mesurement: (qCPR Anne - compression/ventilation feedback software).

SECONDARY OUTCOMES:
Comparison of group A and B: Chest compressions/ventilation ratio | up to 36 months
  Statistic analysis will be used in a comparison of Chest compressions/ventilation ratio in groups A and B.
  Chest compressions/ventilation ratio - good ratio 30:2 according to ERC.
Comparison of group A and B: Depth of chest compressions | up to 36 months
  Statistic analysis will be used to compare the depth of chest compressions in groups A and B.
  Depth of chest compressions: adequate chest compression is 5-6 cm.
Comparison of group A and B: Frequency of chest compression | up to 36 months
  Statistic analysis will be used in a comparison of the frequency of chest compression in groups A and B.
  Frequency of chest compression: adequate average frequency is 100-120/min.
Comparison of group A and B: The longest pause in chest compressions | up to 36 months
  Statistic analysis will be used in a comparison of the longest pause in chest compressions in groups A and B.
  The longest pause in chest compressions: adequate is up to 10s.
Comparison of group A and B: rescue breaths | up to 36 months
  Statistic analysis will be used in a comparison of the longest pause in chest compressions in groups A and B.
  The number of detectable rescue breaths and number of unsuccessful rescue breaths during 2 min in CPR will be statistically analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Martina Kosinová, MD, Study Chair — Masaryk University Faculty of Medicine

IPD SHARING:
Plan to Share IPD: No
The investigators do not plan to share IPD.